CLINICAL TRIAL: NCT05508464
Title: Ablative Radiotherapy to Restrain Every Metastasis Safely Treatable (ARREST-2): A Randomized Phase II/III Trial
Acronym: ARREST2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARREST2; REDA 12529 (Other: London Health Sciences Center Research Institute (LHSCRI))
Record Dates: First submitted 2022-05-13; First posted 2022-08-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard or care palliative radiotherapy (includes the option for no treatment)
  Interventions: Radiation: Arm 1: Standard of Care
- SABR (Active Comparator): SABR to all tumors 6Gy x 5 over 3 weeks
  Interventions: Radiation: Arm 2: SABR

INTERVENTIONS:
Radiation: Arm 2: SABR — SABR to all tumors 6 Gy x 5 over three weeks
  Arms: SABR
Radiation: Arm 1: Standard of Care — Standard of care palliative radiotherapy
  Arms: Standard of Care

SUMMARY:
This is a phase II/III international multicentre randomized trial. Patients will be randomized in a 1:2 ratio between the standard of care (Arm 1) and SABR (Arm 2) to all sites of disease. The study will start as a phase II trial with an opportunity to convert to a phase III trial. The objective of this trial is to determine the impact of SABR on overall survival, progression-free survival, quality of life, and toxicity in patients with polymetastatic disease.

DETAILED DESCRIPTION:
A defining hallmark of cancer is its capability to metastasize. With few exceptions, patients with metastatic disease are considered incurable, and when offered treatment, the intent is to palliate symptoms and delay the inevitable morbidity and mortality that accompanies disease progression. Systemic therapy has been and remains the mainstay of treatment for metastatic disease, however the decision to initiate or continue systemic therapy is a balance of the anticipated benefits and the adverse effects of treatment. Virtually all patients eventually reach a point where systemic therapy will be ceased.

Therapeutic radiotherapy in cancer care can be prescribed with curative or palliative intent. Palliative radiotherapy has long held a role in improving or stabilizing symptoms such as pain, bleeding, or neurologic dysfunction by delivering relatively low radiation doses to metastatic tumours. While palliating symptoms continues to be an important indication, the use of high dose, conformal radiotherapy, termed stereotactic ablative radiotherapy (SABR), has gained traction as an alternative treatment option for select metastatic patients, primarily those with oligometastatic disease.

The objective of this trial is to determine the impact of SABR on overall survival, progression-free survival, quality of life, and toxicity in patients with polymetastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* willing and able to provide informed consent
* ECOG performance status 0-2
* Life expectancy > or equal to 6 months
* Histologically confirmed malignancy with evidence of metastatic disease on imaging
* All sites of disease can be safely treated on a preliminary radiation plan
* > or equal to 11 metastases (the primary tumor does not have to be controlled and can be included as a target if it can feasibly and safely be treated with SABR. If the primary tumor is treated, a minimum of 12 targets are required0 at least 11 metastases are required in addition to the primary tumor.)
* Investigations required within 12 weeks of enrollment:
* Brain: MRI is required for all patients with known untreated or previously treated brain metastases. MRI is strongly recommended for all tumor sites with a propensity to develop brian metastases.
* Body: 18-FDG PET/CT imaging is recommended, except for tumors where FDG uptake is not expected (e.g. prostate, renal cell carcinoma). PSMA-PET or choline-PET is recommended for prostate cancer. In situations where a PET scan is unavailable, or for tumors that do not take up radiotracer, a CT neck/chest/abdomen/pelvis and bone scan are required.
* Liver: For patients with liver metastases, a diagnostic or simulation MRI is required to confirm the total number of metastases.
* No plans for systemic therapy (i.e. chemotherapy, targeted agent, immunotherapy) for 3 months from the time of enrolment. Reasons may include: a break from systemic therapy is desired by the patient and medical oncologist, the patient declines next line of systemic therapy, or no further systemic therapy options are available. Exceptions include hormone therapy for breast cancer or prostate cancer, which may be continued.
* SABR or palliative radiotherapy should commence no later than 2 weeks after randomization.
* For patients with brain metastases that are going to be treated regardless of the study arm, there must be additional extracranial disease present that will be treated with SABR on Arm 2 and not treated with SABR on Arm 1.

Exclusion Criteria:

* Serious medical comorbidities precluding radiotherapy. These include interstitial lung disease in patients requiring thoracic radiation, Chrohn's disease in patients where the GI tract will receive radiotherapy, ulcerative colitis where the bowel will receive radiotherapy and connective tissue disorders such as lupus or scleroderma.
* For patients with liver metastases, moderate/severe liver dysfunction (Child-Pugh B or C)
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy is allowed, as long as the composite plan meets dose constraints herein. For patients treated with radiation previously, biologically effective dose calculations should be used to equate previous doses to the tolerance doses listed in Appendix 1. All such cases must be discussed with the study PI.
* Inability to treat all sites of disease. Any brain metastasis >3 cm in size or a total volume of brain metastases greater than 30 cc.
* Solitary or dominant brian metastasis requiring surgical decompression.
* Radiologic evidence of spinal cord compression.
* Disseminated disease, including leptomeningeal metastases, peritoneal metastases/carcinomatosis, malignant pleural effusion, and lymphangitis carcinomatosis.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Time from randomization to death from any cause, patients followed for 5 years
  Defined as the time form randomization to death from any cause.

SECONDARY OUTCOMES:
Progression-free survival | Time from randomization to disease progression at any disease site, or death. Up to 5 years
  Defined as the time from randomization to disease progression at any site or death.
Quality of life- An individuals perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. | Measured at baseline, then every 3 months from randomization until 2 years, then every 6 months until 5 years.
  Measured using the Functional Assessment of Cancer Therapy: General (FACT-G)
Quality of life- An individuals perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. | Measured at baseline, then every 3 months from randomization until 2 years, then every 6 months until 5 years.
  Measured using the Functional Assessment of Cancer Therapy: EQ-5D-5L
Toxicity of Ablative Radiotherapy | Measured at baseline, on treatment, 6 weeks post treatment, every 3 months from randomization until 2 years, then every 6 months until 5 years.
  Will be assessed using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 5 for each relevant organ site treated.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre- London Regional Cancer Program, London, Ontario, Canada